CLINICAL TRIAL: NCT04042285
Title: Extracorporeal Shockwave Therapy for Diabetic Foot Wounds: A Cohort Study Comparing Extracorporeal Shockwave Therapy to Standard Treatment for Diabetic Foot Wounds
Brief Title: Extracorporeal Shockwave Therapy for Diabetic Foot Wounds
Status: Completed | Type: Observational
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Collaborators: University of Hull (Other)
Responsible Party: Sponsor
Other Study IDs: R2158
Record Dates: First submitted 2019-07-11; First posted 2019-08-01 (Actual); Results first posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-10

CONDITIONS: Diabetic Foot; Wound
Keywords: Diabetic Foot Wound
MeSH Terms: conditions — Diabetic Foot; Wounds and Injuries | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Extracorporeal shockwave therapy: The shockwave therapy will be given at 120 pulses/cm2, penetration 5mm at a dose of 0.1mJ/mm2 at 5 pulses/second (17). Participants will receive 3 sessions of shockwave therapy in a 7-day period. In addition to standard wound care (dressing changes, negative pressure wound therapy, debridement, offloading footwear, glycaemic control and antibiotics, where appropriate).
  Interventions: Device: Extracorporeal shockwave therapy in addition to standard care

INTERVENTIONS:
Device: Extracorporeal shockwave therapy in addition to standard care — Extracorporeal shockwave therapy will be given at 120 pulses/cm2, penetration 5mm at a dose of 0.1mJ/mm2 at 5 pulses/second. Participants will receive 3 sessions of shockwave therapy in a 7-day period. Standard care as per the NICE and IWGDF guidelines.

SUMMARY:
Diabetic wounds post digital amputation have poor healing in 30-45% of cases, resulting in 75% of patients undergoing a further amputation within the year, despite best wound management.

Extracorporeal shockwave therapy is a promising safe and non invasive treatment that has been shown to improve healing in chronic ulcers and burns by promoting healing and decreasing risk of infection.

The study will recruit patients on a hospital ward and outpatient departments who have a diabetic foot wound. Participants will be informed about the study, given an patient information sheet and invited to give informed consent.

Consenting participants will undergo shockwave therapy three times in the seven days after their operation, in addition to standard wound care.

Wound measurements, blood perfusion, tissue integrity, quality of life and pain scores will be recorded at baseline, after the third treatment, 4 weeks, 8 weeks and 12 weeks after recruitment to the study.

The study aims to recruit 25 patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetes mellitus
* Open wound of the foot
* ABPI >0.8
* Age greater than 18 years old
* Able and willing to give written informed consent
* Be able to adhere to protocol and attend all follow up appointments

Exclusion Criteria:

* Pregnancy or breast-feeding
* Current malignancy
* Allergy to materials used in the treatment
* Palliative
* Unable or unwilling to give consent
* Anticoagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic patients with a foot wound
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-02-02 (Actual); Study Completion 2022-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George E Smith, M.D, Principal Investigator — Academic Vascular Surgery Unit
Locations (1):
- Hull and East Yorkshire Hospitals NHS Trust, Hull, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Extracorporeal Shockwave Therapy: The shockwave therapy will be given at 120 pulses/cm2, penetration 5mm at a dose of 0.1mJ/mm2 at 5 pulses/second (17). Participants will receive 3 sessions of shockwave therapy in a 7-day period. In addition to standard wound care (dressing changes, negative pressure wound therapy, debridement, offloading footwear, glycaemic control and antibiotics, where appropriate).
  Extracorporeal shockwave therapy: Extracorporeal shockwave therapy will be given at 120 pulses/cm2, penetration 5mm at a dose of 0.1mJ/mm2 at 5 pulses/second. Participants will receive 3 sessions of shockwave therapy in a 7-day period.
Period: Overall Study
Arm/Group | Extracorporeal Shockwave Therapy
Started | 24
Completed | 18
Not Completed | 6

BASELINE CHARACTERISTICS:
Population: These are patients with a diabetic foot wound who meet the eligibility criteria.
Arm/Group | Extracorporeal Shockwave Therapy
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.82 (13.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 24
Wound Volume [Median (Standard Deviation); unit: mm^3] | 1071.14 (1416.56)

OUTCOME MEASURES:

1. Primary Outcome: Wound Volume
Description: Change in wound volume between study visits
Time Frame: 12 weeks
Measure: Mean (95% Confidence Interval); unit: cm^3
Arm/Group | Extracorporeal Shockwave Therapy
Number analyzed (Participants) | 22
cm^3 | 1.16 [-1.8 to 4.12]

2. Secondary Outcome: Pain Questionnaire
Description: Brief Pain Inventory (BPI) - A person rates their pain on a scale of 0 to 10. The BPI scale defines pain as follows: Worst Pain Score: 1 - 4 = Mild Pain. Worst Pain Score: 5 - 6 = Moderate Pain. Worst Pain Score: 7 - 10 = Severe Pain.
Time Frame: 12 weeks
Measure: Median (Standard Deviation); unit: Score on a scale
Arm/Group | Extracorporeal Shockwave Therapy
Number analyzed (Participants) | 24
Score on a scale | 1 (0)

3. Secondary Outcome: Quality of Life Questionnaires SF-12
Description: Quality of Life Questionnaire Short Form-12 (8 domains of questions) scored on a scale 1-5, where a low score is good health and a high score is poor health. Total scores range from 0 to100, with higher scores indicating better physical and mental health functioning.
Time Frame: 12 weeks
Measure: Median (Standard Deviation); unit: Score on scale
Arm/Group | Extracorporeal Shockwave Therapy
Number analyzed (Participants) | 24
Score on scale | 59.78 (6.13)

4. Secondary Outcome: Infection Rate
Description: The number of wounds which develop an infection in the study period.
Time Frame: Recorded at 12 weeks
Measure: Number; unit: Infection that developed per ulcer
Units Other Than Participants: Ulcers
Arm/Group | Extracorporeal Shockwave Therapy
Number analyzed (Participants) | 24
Number analyzed (Ulcers) | 24
Infection that developed per ulcer | 1

5. Secondary Outcome: Minor Amputation Rate
Description: The number of minor amputations of treated limbs in the study period.
Time Frame: Recorded at 12 weeks
Measure: Number; unit: Index limb
Units Other Than Participants: Index limb
Arm/Group | Extracorporeal Shockwave Therapy
Number analyzed (Participants) | 24
Number analyzed (Index limb) | 24
Index limb | 2

6. Secondary Outcome: Local Perfusion Rate
Description: Blood flow perfusion rate of superficial tissues using Doppler flowmetry, an increase in the number signifies an increase in bloodflow to the area. Doppler flowmetry measures the shift in frequency that occurs when light is scattered by the red blood cells moving through capillaries.
Time Frame: 7 days
Measure: Median (Standard Deviation); unit: ml/ml/s
Arm/Group | Extracorporeal Shockwave Therapy
Number analyzed (Participants) | 24
ml/ml/s | 28.85 (37.09)

7. Secondary Outcome: Tissue Integrity
Description: Tissue hydration determined by a vapometer, the sensor evaluates the efficiency of the human skin water barrier, a high score is a sign of increased tissue water loss, and therefore reduced tissue integrity.
Time Frame: 7 days
Measure: Median (Standard Deviation); unit: g/m^2h
Arm/Group | Extracorporeal Shockwave Therapy
Number analyzed (Participants) | 24
g/m^2h | 21.53 (12.93)

8. Secondary Outcome: Quality of Life Questionnaire EQ5D3L
Description: The EuroQoL-5D-5L is a brief, multiattribute, generic, health status measure composed of 5 questions with Likert response options. EQ-5D-5L index scores range from -0.59 to 1, where 1 is the best possible health state.
Time Frame: 12 weeks
Measure: Median (Standard Deviation); unit: Score on a scale
Arm/Group | Extracorporeal Shockwave Therapy
Number analyzed (Participants) | 24
Score on a scale | 0.81 (0.44)

ADVERSE EVENTS:
Time Frame: 12 week adverse event rate.
Arm/Group | Extracorporeal Shockwave Therapy
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-01): https://cdn.clinicaltrials.gov/large-docs/85/NCT04042285/Prot_SAP_000.pdf